CLINICAL TRIAL: NCT04081792
Title: Optimization of the Surgical and Medical Management of Diabetic Foot Infections
Brief Title: Optimal Antibiotics for Operated Diabetic Foot Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFI_Cohort
Record Dates: First submitted 2019-08-05; First posted 2019-09-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot Infection; Surgical Wound; Antibiotic Side Effect; Infection
Keywords: diabetic foot; osteomyelitis; amputation; antibiotics
MeSH Terms: conditions — Surgical Wound; Infections; Diabetic Foot; Osteomyelitis | interventions — Anti-Infective Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- 1. Trial (Amputation) Soft tissue - short antibiotic arm (Experimental): The intervention group consists of 1 day of postoperative antibiotic therapy for eventual residual soft tissue infection after amputation.
  Interventions: Procedure: Antibiotic therapy
- 1. Trial (Amputation) Soft tissue - long antibiotic arm (Active Comparator): The control group consists of 4 days duration of postoperative antibiotic therapy for eventual residual soft tissue infection after amputation.
  Interventions: Procedure: Antibiotic therapy
- 1. Trial (Amputation) Bone - short antibiotic arm (Experimental): The intervention group consists of 1 week of postoperative antibiotic therapy for eventual residual bone infection / contamination in the proximal bone stump after amputation.
  Interventions: Procedure: Antibiotic therapy
- 1. Trial (Amputation) Bone - long antibiotic arm (Active Comparator): The intervention group consists of 3 weeks of postoperative antibiotic therapy for eventual residual bone infection / contamination in the proximal bone stump after amputation.
  Interventions: Procedure: Antibiotic therapy
- 2.Trial (soft tissue infection) - short antibiotic arm (Experimental): The intervention group consists of 10 days of post-debridement antibiotic therapy for non-amputated diabetic foot soft tissue infection.
  Interventions: Procedure: Antibiotic therapy
- 2. Trial (soft tissue infection) - long antibiotic arm (Active Comparator): The control group consists of 20 days of post-debridement antibiotic therapy for non-amputated diabetic foot soft tissue infection.
  Interventions: Procedure: Antibiotic therapy
- 2. Trial (osteomyelitis) - short antibiotic arm (Experimental): The intervention group consists of 3 weeks of post-debridement antibiotic therapy for non-amputated diabetic foot osteomyelitis.
  Interventions: Procedure: Antibiotic therapy
- 2. Trial (osteomyelitis) - long antibiotic arm (Active Comparator): The control group consists of 6 weeks of post-debridement antibiotic therapy for non-amputated diabetic foot osteomyelitis.
  Interventions: Procedure: Antibiotic therapy

INTERVENTIONS:
Procedure: Antibiotic therapy — Postoperative randomizations regarding the duration of systemic antibiotics

SUMMARY:
Diabetic foot problems, especially infections (DFI), require multiple resources including iterative surgeries and amputations, long-lasting antibiotic therapies, education, off-loading and eventually revascularization and appropriate foot-ware. Treatment is complicated, multidisciplinary, and marked with a high risk of recurrences.

This is a retrospective and prospective cohort with side studies of pathologies and academic research questions that cannot be separated from each other.

The investigators establish a retro-and prospective cohort of diabetic foot problems (ambulatory and hospitalized patients) and perform side studies to reduce the incidence of complications, and to reduce recurrences of DFI, cost and adverse events related to therapies.

Cohort: Prospective and retrospective cohort of all diabetic foot problems with emphasis on surgical and infectious variables.

Trial 1 (Randomized trial on residual infection after amputation):

Determination of the level of amputation per MRI followed by a randomization concerning the duration of post-amputation systemic antibiotic therapy, if there is residual bone infection.

Trial 2 (Randomized trial on infection without amputation):

Determination of the duration of systemic antibiotic therapy in diabetic foot infections without Amputation of the infection.

DETAILED DESCRIPTION:
Trial 1: At enrollment (Day 1), the investigator will prescribe empiric antibiotic treatment based on instructions provided in the protocol and determine the most appropriate route of administration (oral or IV) according to the patient's condition. Patients will be randomized in the ratio 1:1 between 1 versus 4 days for post-amputation soft tissue infections; and between 1 versus 3 weeks if there is microbiologically proven residual bone infection/contamination in the proximal stump samples of the residual bone.

Trial 2: At enrollment (Day 1), the investigator will prescribe empiric antibiotic treatment based on instructions provided in the protocol and determine the most appropriate route of administration (oral or IV) according to the patient's condition. Patients will be randomized in the ratio 1:1 between 10 versus 20 days for post-debridement soft tissue infections; and between 3 versus 6 weeks for diabetic foot osteomyelitis post.-debridement (without amputation).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diabetic foot infections or ischemia/necrosis with surgical amputation/disarticulation level in vicinity of MRI signs of infection
* At least two months of follow-up from hospitalization
* Patient signing to participate, including acceptance of local wound care, -off-loading and arterial re-vascularization (if clinically indicated).

Exclusion Criteria:

* At least 5 cm of distance between amputation level and infection.
* Any concomitant infection requiring more than 5 days of systemic antibiotic therapy
* Eventual osteosynthesis material not removed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a clinical and microbiological remission of treated infection at 2 months | Through study completion, at 2 months
  Remission is the absence of any anamnesis or clinics for persistent or recurrent infection

SECONDARY OUTCOMES:
Anatomical Amputation Level Determination by MRI | At study entry, Day O
  Evaluation of the accuracy of the extension of infection. Surgical decision for amputation level per magnetic resonance imaging when compared to microbiology, histology and intraoperative assessment.
Rates of adverse events of antibiotic therapy | Through study completion, at 2 months
  Outcome of antibiotic-related adverse events
Duration of wound healing time | Through study completion, at 2 months
  Evolution of wound size under therapy and off-loading over time. Wound Score.
Numbers of Cost and resource reductions | Through study completion, at 2 months
  Overall hospitalization and treatment costs; in Swiss Francs
Scales of Patient's satisfaction | Through study completion, at 2 months
  Questionnaires and Scores (e.g. AOFAS Score) ranging from 0 to 1. Alternatively, a home made Likert Scale ranging from 0 to 7 Points will be used.
Statistical evaluation of risk factors for failure of remission | 2 years
  Multivariate Cox Regression analyses

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, PD MD, Study Director — Balgrist University Hospital, Zurich, Switzerland
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
not yet determined in detail
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: In 2022
Access Criteria: Upon reasonable request upon the contact authors

REFERENCES:
- [Background] Uckay I, Jornayvaz FR, Lebowitz D, Gastaldi G, Gariani K, Lipsky BA. An Overview on Diabetic Foot Infections, including Issues Related to Associated Pain, Hyperglycemia and Limb Ischemia. Curr Pharm Des. 2018;24(12):1243-1254. doi: 10.2174/1381612824666180302145754. PMID 29508677
- [Background] Coster MC, Rosengren BE, Bremander A, Brudin L, Karlsson MK. Comparison of the Self-reported Foot and Ankle Score (SEFAS) and the American Orthopedic Foot and Ankle Society Score (AOFAS). Foot Ankle Int. 2014 Oct;35(10):1031-6. doi: 10.1177/1071100714543647. Epub 2014 Jul 11. PMID 25015390
- [Result] Rossel A, Lebowitz D, Gariani K, Abbas M, Kressmann B, Assal M, Tscholl P, Stafylakis D, Uckay I. Stopping antibiotics after surgical amputation in diabetic foot and ankle infections-A daily practice cohort. Endocrinol Diabetes Metab. 2019 Feb 6;2(2):e00059. doi: 10.1002/edm2.59. eCollection 2019 Apr. PMID 31008367
- [Result] Uckay I, Berli M, Sendi P, Lipsky BA. Principles and practice of antibiotic stewardship in the management of diabetic foot infections. Curr Opin Infect Dis. 2019 Apr;32(2):95-101. doi: 10.1097/QCO.0000000000000530. PMID 30664029
- [Result] Gariani K, Lebowitz D, von Dach E, Kressmann B, Lipsky BA, Uckay I. Remission in diabetic foot infections: Duration of antibiotic therapy and other possible associated factors. Diabetes Obes Metab. 2019 Feb;21(2):244-251. doi: 10.1111/dom.13507. Epub 2018 Sep 21. PMID 30129109
- [Derived] Zendeli F, Jedrusik A, Schaefer RO, Albrecht D, Betz M, Waibel FWA, Grober T, Kuhne N, Konneker S, Uckay I. Pathogen-Specific Risk for Iterative Surgical Debridement in Orthopedic Infections: A Prospective Multicohort Analysis. J Clin Med. 2025 Dec 10;14(24):8750. doi: 10.3390/jcm14248750. PMID 41464652
- [Derived] Waibel F, Berli M, Catanzaro S, Sairanen K, Schoni M, Boni T, Burkhard J, Holy D, Huber T, Bertram M, Laubli K, Frustaci D, Rosskopf A, Botter S, Uckay I. Optimization of the antibiotic management of diabetic foot infections: protocol for two randomized controlled trials. Trials. 2020 Jan 8;21(1):54. doi: 10.1186/s13063-019-4006-z. PMID 31915048

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT04081792/SAP_000.pdf